CLINICAL TRIAL: NCT00896675
Title: Proteomic Prediction of Clinical Benefit in HNSCC
Brief Title: Blood Proteins in Predicting Treatment Benefit in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0744; P30CA068485 (NIH); VU-VICC-HN-0744; VU-VICC-070359
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage IV salivary gland cancer; recurrent salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients treated with EGFR inhibitors and/or VEGF inhibitor
  Interventions: Other: proteomic profiles
- NOT treated with EGFR inhibitors and/or VEGF inhibitor
  Interventions: Other: proteomic profiles

INTERVENTIONS:
Other: proteomic profiles — blood samples analysis
  Groups: patients treated with EGFR inhibitors and/or VEGF inhibitor
Other: proteomic profiles — blood samples analysis
  Groups: NOT treated with EGFR inhibitors and/or VEGF inhibitor

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory may help doctors learn more about cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at proteins in blood samples to predict treatment benefit in patients with recurrent and/or metastatic squamous cell head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify head and neck squamous cell cancer patients who will benefit from treatment with the EGFR inhibitors (i.e., erlotinib hydrochloride, gefitinib, and cetuximab) and VEGF inhibitor (i.e., bevacizumab), based on predictive proteomic profiles in patient blood samples.

OUTLINE: This is a multicenter study.

Blood samples are analyzed for proteomic profile to determine good and bad prognoses in patients treated with or without EGFR inhibitors and/or a VEGF inhibitor.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell head and neck cancer

  * Recurrent and/or metastatic disease
* Meets 1 of the following criteria:

  * Previously treated with EGFR inhibitors and/or VEGF inhibitor on 1 of the following clinical trials, and has available blood samples:

    * A Phase I/II Study of Bevacizumab (rhu MAb VEGF) in Combination With OSI-774 for Patients With Recurrent or Metastatic Cancer of the Head and Neck
    * A Phase II Study of 250-mg ZD1839 Monotherapy in Recurrent or Metastatic or Both Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck
  * Previously treated with cetuximab and has blood samples available from protocol VU-VICC-HN-0356
  * Previously treated with conventional chemotherapy and has blood samples available from protocol VU-VICC-HN-0356

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head and Neck cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Identification of patients who will benefit from treatment with EGFR and/or VEGF inhibitors based on serum proteomic profiles | upon analysis of each patient tissue collection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee